CLINICAL TRIAL: NCT06664645
Title: Evaluation of Rotator Cuff Repair With Long Head of the Biceps Reinforcement: a Prospective Randomized Study
Brief Title: Rotator Cuff Tears Treated With Long Head of the Biceps Reinforcement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Responsible Party: Principal Investigator, GUSTAVO DE MELLO RIBEIRO PINTO, Principal investigator, Hospital Universitario Pedro Ernesto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 53239121.4.0000.5259
Record Dates: First submitted 2024-10-11; First posted 2024-10-29 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Rotator Cuff Injuries; Biceps Tendon Reattachment
Keywords: rotator cuff; tendon transfer; biceps reinforcement; biceps autograft
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: A prospective randomized study will be carried out in a 1:1 ratio between groups. Patients with large and extensive rotator cuff injuries will be selected at the Shoulder and Elbow clinic of Pedro Ernesto University Hospital (HUPE-UERJ), during outpatient care.
  Patients with an intact long head of the biceps will be randomized into two groups, according to the use or not of the tendon: complete repair with LHB tendon reinforcement and complete repair without reinforcement.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- complete repair with LHB tendon reinforcement (Experimental): complete repair with LHB tendon reinforcement
  Interventions: Procedure: LHB tendon reinforcement
- complete repair without reinforcement (Active Comparator): complete repair without reinforcement.
  Interventions: Procedure: complete repair without reinforcement

INTERVENTIONS:
Procedure: LHB tendon reinforcement — complete repair with LHB tendon reinforcement
  Arms: complete repair with LHB tendon reinforcement
Procedure: complete repair without reinforcement — conventional rotator cuff complete repair without reinforcement
  Arms: complete repair without reinforcement

SUMMARY:
The increase of the population life expectancy and the active lifestyle adopted in recent years have contributed to the higher incidence of rotator cuff injuries. For large (>3 cm) and extensive (>5 cm) injuries of the rotator cuff, even after complete or partial repair, the chances of failure reach 94%.

An alternative in rotator cuff injuries is the use of the long head of the biceps (LHB) as an autologous graft to increase the healing rate and the final outcomes.

The primary objective is to compare the functional results, according to the ASES score, between patients who use or not the long head biceps brace for complete repairs of large and extensive rotator cuff tears.

The secondary objectives are to compare the groups according to structural results by MRI and functional results by the UCLA score.

DETAILED DESCRIPTION:
A prospective randomized study will be carried out in a 1:1 ratio between groups. Patients with large and extensive rotator cuff injuries will be selected at the Shoulder and Elbow clinic of Pedro Ernesto University Hospital (HUPE-UERJ), during outpatient care.

Patients with an intact long head of the biceps will be randomized into two groups, according to the use or not of the tendon: complete repair with LHB tendon reinforcement and complete repair without reinforcement. All patients will be operated by the same surgeon.

All selected patients will be explained what the research is about by a research assistant not involved in the treatment and will be offered the option to participate or not.

The "American Shoulder and Elbow Surgeons Standardized Shoulder Assessment Form" (ASES) scale will be adopted as the primary outcome. The "Modified University of California at Los Angeles Shoulder Rating Scale" (UCLA) and the assessment of tendon healing with magnetic resonance imaging at 6 months after surgery, using the classification of Sugaya et al. will be secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Long head tendon of biceps intact;
* Large or extensive posterosuperior rotator cuff injuries according to the classification of DeOrio and Cofield;20
* Fatty degeneration of the ≦2 supraspinatus muscle according to the classification of Goutallier.21

Exclusion Criteria:

* Active or previous infection in the affected shoulder;
* Patients unable to understand preoperative questionnaires;
* Patient who does not undergo at least 1 postoperative evaluation.
* Injury where complete repair of the rotator cuff is not possible;
* Rupture of the LHB tendon diagnosed intraoperatively.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Visual analogue score (VAS) | 24 months
  Visual analogue score: it is a 10 cm line with two end points, one representing "no pain" and the other representing "worst pain". The patient marks the line to indicate their current pain level, and the distance from the "no pain" marker to the mark is measured in centimeters to provide a score. A higher score indicates greater pain intensity.
Structural outcomes | 24 months
  Patients will undergo preoperative MRI and from 6 months after the procedure. All images will be evaluated by at least two authors of the work, who will not know which group the patients belong to.
  The classification by Sugaya et al. stratifies the appearance of the tendon after repair into 5 types: type I (sufficient thickness with low signal in all images); type II (sufficiently thick with high focal signal); type III (insufficient thickness without discontinuity); type IV (small size tear) and type V (medium or large size tear).
  The healing of the long head biceps reinforcement will also be evaluated by MRI and classified as unhealed and healed.
American Shoulder and Elbow Score (ASES) | 24
  American Shoulder and Elbow Score score ranges from 0 to 100, with 0 the lowest level of function and 100 the highest level of function.
The University of California-Los Angeles (UCLA) | 24 months
  Scores ranged from 0 to 35 with a score of 0 indicating worst shoulder function and 35 indicating best shoulder function.
The 12 item Short Form Survey (SF-12) | 24 months
  This is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  Utilize the norm-based scoring system to interpret Physical component and Mental component scores, with a mean of 50 and a standard deviation of 10 in the general population. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.

CONTACTS AND LOCATIONS:
Locations (1):
- hospital Universitário Pedro Ernesto, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barth J, Olmos MI, Swan J, Barthelemy R, Delsol P, Boutsiadis A. Superior Capsular Reconstruction With the Long Head of the Biceps Autograft Prevents Infraspinatus Retear in Massive Posterosuperior Retracted Rotator Cuff Tears. Am J Sports Med. 2020 May;48(6):1430-1438. doi: 10.1177/0363546520912220. Epub 2020 Apr 8. PMID 32267730
- [Background] Rhee SM, Youn SM, Park JH, Rhee YG. Biceps Rerouting for Semirigid Large-to-Massive Rotator Cuff Tears. Arthroscopy. 2021 Sep;37(9):2769-2779. doi: 10.1016/j.arthro.2021.04.008. Epub 2021 Apr 20. PMID 33892075
- [Background] Cho NS, Yi JW, Rhee YG. Arthroscopic biceps augmentation for avoiding undue tension in repair of massive rotator cuff tears. Arthroscopy. 2009 Feb;25(2):183-91. doi: 10.1016/j.arthro.2008.09.012. Epub 2008 Nov 1. PMID 19171279